CLINICAL TRIAL: NCT01120899
Title: A Pilot Study for the Evaluation of Minocycline as a Microglia Inhibitor in the Treatment of Diabetic Macular Edema
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Collaborators: The Emmes Company, LLC (Industry)
Responsible Party: Principal Investigator, Catherine Cukras, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 100098; 10-EI-0098 (Other: CNS IRB)
Record Dates: First submitted 2010-05-08; First posted 2010-05-11 (Estimated); Results first posted 2012-09-06 (Estimated); Last update posted 2014-10-17 (Estimated); Status verified 2014-10

CONDITIONS: Diabetic Macular Edema
Keywords: Diabetic Macular Edema; Microglia; Minocycline; Diabetes
MeSH Terms: conditions — cyclopia sequence; Diabetes Mellitus | interventions — Minocycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Minocycline (Experimental)
  Interventions: Drug: Minocycline

INTERVENTIONS:
Drug: Minocycline — Participants take 100 mg minocycline pills twice daily for 24 months.
  Other Names: Dynacin; serial number 73419626; Minocin; serial number 72309825; Minocin PAC; Myrac; serial number 76589055; Solodyn; serial number 78883462; Vectrin; serial number 78188505

SUMMARY:
The objective of this study is to investigate the safety and efficacy of minocycline as a microglia inhibitor in individuals with diabetic macular edema (DME).

DETAILED DESCRIPTION:
Objective: Diabetic retinopathy (DR) is one of the leading causes of blindness in the United States. A frequent manifestation of diabetic retinopathy is diabetic macular edema (DME) for which the only proven treatment is laser photocoagulation. In the retina, microglia are capable of migrating through the retina to sites of inflammation to associate closely with neurons and the vasculature, and are key cellular players in the mediation of processes of chronic inflammation implicated in DME. For these reasons, microglia represent a promising cellular target for forms of therapy that limit the deleterious inflammatory changes found in DR. The objective of this study is to investigate the safety and efficacy of minocycline as a microglia inhibitor in patients with DME.

Study Population: Eligibility criteria include previous treatment with standard-of-care focal laser photocoagulation, or macular edema not amenable to focal laser treatment; retinal thickness in the central subfield > 250 microns as measured by optical coherence tomography (OCT); and visual acuity between 20/32 and 20/200 in the study eye.

Design: Five participants will be initially enrolled in this open-label pilot study. However, up to an additional three participants may be enrolled to account for participants who withdraw from the study prior to receipt of six months of study treatment. Participants will take an oral dose of 100 mg of minocycline twice daily for 24 months. During each visit, participants will have their visual acuity measured and will undergo OCT testing to measure retinal thickness. Beginning at the Month 6 visit, participants will be eligible for focal laser therapy unless they show marked improvement in retinal thickness and/or visual acuity or if they are not amenable to focal laser treatment. Participants who do not meet the criteria for improvement will also be eligible for anti-vascular endothelial growth factor (VEGF) treatments such as bevacizumab (Avastin®) or ranibizumab (Lucentis®). Additionally, beginning at the Month 4 visit, participants will be assessed for worsening disease defined as loss of ≥ 15 Early Treatment Diabetic Retinopathy Study (ETDRS) letters of vision compared to baseline or a ≥ 50% increase in total retinal thickness as measured by OCT. Participants deemed to have worsening disease will also be eligible for focal laser and/or anti-VEGF treatments.

Outcome Measures: The primary outcome is the change in best-corrected visual acuity (BCVA) in the study eye at 6 months compared to baseline. Secondary outcomes include the change in retinal thickness as measured by OCT at 6, 12, 18 and 24 months compared to baseline, change in BCVA at 12, 18 and 24 months compared to baseline, as well as changes in fluid leakage in the macula as demonstrated by fluorescein angiography at 6, 12, 18 and 24 months compared to baseline. Safety outcomes include the number and severity of systemic and ocular toxicities, and adverse events.

ELIGIBILITY:
Inclusion Criteria

1. Participant is 18 years of age or older.
2. Participant must understand and sign the protocol's informed consent document.
3. Female participants of childbearing potential (see Appendix 1 for definition) must not be pregnant or breast-feeding, must have a negative urine pregnancy test within 24 hours prior to initiation of study medication and must be willing to undergo urine pregnancy tests throughout the study.
4. Female participants of childbearing potential (see Appendix 1 for definition) and male participants able to father children must have (or have a partner who has) had a hysterectomy or vasectomy, be completely abstinent from intercourse or must agree to practice two acceptable methods of contraception throughout the course of the study and for one week after study medication discontinuation (based on the half life of minocycline which is 11-22 hours). Acceptable methods of contraception include:

   * hormonal contraception (i.e., birth control pills*, injected hormones, dermal patch or vaginal ring),
   * intrauterine device,
   * barrier methods (diaphragm, condom) with spermicide, or
   * surgical sterilization (hysterectomy or tubal ligation). *Oral birth control pills must be used with caution as minocycline decreases the effectiveness of some oral contraceptives. Participants already taking oral contraceptives may continue to use them, but must agree to use at least one other method of birth control while on study.
5. Participants must agree to notify the study investigator or coordinator if any of their doctors initiate a new medication during the course of this study.
6. Participant must have normal renal function and liver function or have mild abnormalities no greater than grade 1 as defined by the Common Terminology Criteria for Adverse Events v4.0 (CTCAE). Refer to Appendix 2 for grading.
7. Participant has a diagnosis of diabetic mellitus (type 1 or type 2). Any one of the following will be considered to be sufficient evidence that diabetes is present:

   * Current regular use of insulin for the treatment of diabetes
   * Current regular use of oral anti-hyperglycemia agents for the treatment of diabetes
   * Documented diabetes by American Diabetes Association (ADA) and/or World Health Organization (WHO) criteria
8. Participant has documented hemoglobin A1C 12% or less within one month of baseline.
9. Participant must agree to minimize exposure to sunlight or artificial UV rays and to wear protective clothing, sunglasses and sunscreen [minimum Sun Protection Factor (SPF) 15] if s/he must be out in the sun.
10. Participant has at least one eye that meets the study eye criteria listed below.

Exclusion Criteria

1. Participant is in another investigational study and actively receiving study therapy.
2. Participant is unable to comply with study procedures or follow-up visits.
3. Participant has a known hypersensitivity to sodium fluorescein dye.
4. Participant has a condition that, in the opinion of the investigator, would preclude participation in the study (e.g., unstable medical status including blood pressure and glycemic control).

   • Patients in poor glycemic control who, within the last four months, initiated intensive insulin treatment (a pump or multiple daily injections) or plan to do so in the next four months should not be enrolled.
5. Participant has a history of chronic renal failure requiring dialysis or kidney transplant.
6. Participant has a history of hepatitis or liver failure.
7. Participant has an allergy or hypersensitivity to minocycline or any drug in the tetracycline family.
8. Participant is taking any medication that could adversely interact with minocycline such as methoxyflurane.
9. Participant has a blood pressure of > 180/110 (systolic above 180 OR diastolic above 110).

   • If blood pressure is brought below 180/110 by anti-hypertensive treatment, patient can become eligible.
10. Participant has a history of treatment with systemic anti-vascular endothelial growth factor (VEGF) agents or steroids within three months prior to study entry.
11. Participant has a history of thyroid cancer.

Study Eye Inclusion Criteria

1. Best-corrected Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity score between 78 and 39 letters (i.e., between 20/32 and 20/200).
2. Definite retinal thickening due to diabetic macular edema based on clinical exam involving the center of the macula that is not refractory to further therapy as based on the investigator's clinical judgment.
3. Previous treatment with focal laser photocoagulation following standard-of-care/best practice guidelines, as described by the ETDRS study,6 ≥ 3 months prior to enrollment unless the edema is not responsive to previous laser and/or not amenable to safe laser treatment at the discretion of the investigator. The laser treatment may be performed at the National Eye Institute (NEI) clinical center (CC) or by an outside ophthalmologist at the discretion of the participant and the investigator.
4. Retinal thickness in the central subfield on baseline optical coherence tomography (OCT) measurement > 250 microns, as measured by Spectral OCT.
5. Media clarity, pupillary dilation and patient cooperation sufficient for adequate fundus photographs.

Study Eye Exclusion Criteria

1. Macular edema is considered to be due to a cause other than diabetic macular edema.

   An eye should not be considered eligible if:
   * The macular edema is considered to be related to cataract extraction or
   * Clinical exam and/or OCT suggest that vitreoretinal interface disease (e.g., a taut posterior hyaloid or epiretinal membrane) is the primary cause of the macular edema.
2. An ocular condition is present such that, in the opinion of the investigator, visual acuity would not improve from resolution of macular edema (e.g., foveal atrophy, pigmentary changes, dense subfoveal hard exudates, non-retinal condition).
3. An ocular condition is present (other than diabetic retinopathy) that, in the opinion of the investigator, might affect macular edema or alter visual acuity during the course of the study (e.g., vein occlusion, uveitis or other ocular inflammatory disease, neovascular glaucoma, Irvine-Gass Syndrome, etc.).
4. Substantial cataract that, in the opinion of the investigator, is likely to be decreasing visual acuity by three lines or more (i.e., cataract would be reducing acuity to 20/40 or worse if eye was otherwise normal).
5. History of panretinal scatter photocoagulation (PRP) within four months prior to study entry.
6. History of prior pars plana vitrectomy within six months prior to study entry.
7. History of major ocular surgery (including cataract extraction, scleral buckle, any intraocular surgery, etc.) within three months prior to study entry.
8. History of yttrium aluminium garnet (YAG) capsulotomy performed within two months prior to study entry.
9. History of treatment within three months prior to enrollment with any drug that has not received regulatory approval at the time of study entry, such as intravitreal or periocular steroids or intravitreal anti-VEGF agents.

Choice of Study Eye in Cases of Bilateral Disease

If both eyes of a participant meet the study eye inclusion and exclusion criteria listed above, the following will be used to determine the study eye:

1. If one eye is treatment-naïve and the other is not, the treatment-naïve eye will be chosen as the study eye.
2. If both eyes are treatment-naïve, the eye with the better visual acuity will be chosen as the study eye.
3. If both eyes are treatment-naïve and are equivalent, the choice of study eye will be determined at the investigator's discretion after consultation with the participant.
4. If both eyes have been previously treated, the choice of study eye will be determined at the investigator's discretion after consultation with the participant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2010-04; Primary Completion 2011-08 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine A Cukras, MD, PhD, Principal Investigator — National Eye Institute (NEI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Kempen JH, O'Colmain BJ, Leske MC, Haffner SM, Klein R, Moss SE, Taylor HR, Hamman RF; Eye Diseases Prevalence Research Group. The prevalence of diabetic retinopathy among adults in the United States. Arch Ophthalmol. 2004 Apr;122(4):552-63. doi: 10.1001/archopht.122.4.552. PMID 15078674
- [Background] Klein R, Klein BE, Moss SE, Davis MD, DeMets DL. The Wisconsin epidemiologic study of diabetic retinopathy. IV. Diabetic macular edema. Ophthalmology. 1984 Dec;91(12):1464-74. doi: 10.1016/s0161-6420(84)34102-1. PMID 6521986
- [Background] Ferris FL 3rd, Patz A. Macular edema: a major complication of diabetic retinopathy. Trans New Orleans Acad Ophthalmol. 1983;31:307-16. No abstract available. PMID 6623578
- [Result] Cukras CA, Petrou P, Chew EY, Meyerle CB, Wong WT. Oral minocycline for the treatment of diabetic macular edema (DME): results of a phase I/II clinical study. Invest Ophthalmol Vis Sci. 2012 Jun 22;53(7):3865-74. doi: 10.1167/iovs.11-9413. PMID 22589436
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2010-EI-0098.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Minocycline: Participants take an oral dose of 100 mg of minocycline twice daily for 24 months.
Period: Overall Study
Arm/Group | Minocycline
Started | 6
Month 6 | 5
Month 12 | 3
Month 18 | 3
Completed | 3
Not Completed | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | Minocycline
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.8 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Secondary Outcome: Change in BCVA in the Study Eye at 6 Months Compared to Baseline
Description: Visual acuity was measured using the Early Treatment Diabetic Retinopathy Study (ETDRS) protocol. Acuity is measured as letters read on an ETDRS eye chart and the letters read equate to Snellen measurements. For example, if a participant reads between 84 and 88 letters, the equivalent Snellen measurement is 20/20.
  The participant's eye that met the study eye eligibility criteria was selected as the study eye. For cases in which both eyes met the study eye eligibility criteria, the study eye was selected according to the "choice of study eye in cases of bilateral disease" selection criteria outlined in the eligibility criteria. The eye not chosen as the study eye is referred to as the "fellow eye."
Time Frame: Baseline and 6 Months
Measure: Mean (Standard Deviation); unit: ETDRS Letters
Units Other Than Participants: Eyes
Arm/Group | Minocycline
Number analyzed (Participants) | 5
Number analyzed (Eyes) | 5
ETDRS Letters | 5.8 (5.4)

2. Secondary Outcome: Change in BCVA in the Study Eye at 12 Months Compared to Baseline
Description: as for outcome 1
Time Frame: Baseline and 12 Months
Measure: Mean (Standard Deviation); unit: ETDRS Letters
Units Other Than Participants: Eyes
Arm/Group | Minocycline
Number analyzed (Participants) | 3
Number analyzed (Eyes) | 3
ETDRS Letters | 8.0 (8.9)

3. Secondary Outcome: Change in BCVA in the Study Eye at 18 Months Compared to Baseline
Description: Visual acuity was measured using the Early Treatment Diabetic Retinopathy Study (ETDRS) protocol. Acuity is measured as letters read on an ETDRS eye chart and the letters read equate to Snellen measurements. For example, if a participant reads between 84 and 88 letters, the equivalent Snellen measurement is 20/20.
Time Frame: Baseline and 18 Months
Measure: Mean (Standard Deviation); unit: ETDRS letters
Units Other Than Participants: Eyes
Arm/Group | Minocycline
Number analyzed (Participants) | 3
Number analyzed (Eyes) | 3
ETDRS letters | 9.0 (4.0)

4. Secondary Outcome: Change in BCVA in the Study Eye at 24 Months Compared to Baseline
Description: as for outcome 3
Time Frame: Baseline and 24 Months
Measure: Mean (Standard Deviation); unit: ETDRS letters
Units Other Than Participants: Eyes
Arm/Group | Minocycline
Number analyzed (Participants) | 3
Number analyzed (Eyes) | 3
ETDRS letters | 9.3 (6.8)

5. Secondary Outcome: Percentage Change in Retinal Thickness in the Study Eye at 6 Months Compared to Baseline
Description: Retinal thickness was assessed by spectral-domain optical coherence tomography (Cirrus HD-OCT; Carl Zeiss Meditec, Dublin, CA), a non-invasive imaging technique that uses long-wavelength light to capture micrometer-resolution cross-sectional images from biological tissue.
  The participant's eye that met the study eye eligibility criteria was selected as the study eye. For cases in which both eyes met the study eye eligibility criteria, the study eye was selected according to the "choice of study eye in cases of bilateral disease" selection criteria outlined in the eligibility criteria. The eye not chosen as the study eye is referred to as the "fellow eye."
Time Frame: Baseline and 6 Months
Measure: Mean (Standard Deviation); unit: percentage change
Units Other Than Participants: Eyes
Arm/Group | Minocycline
Number analyzed (Participants) | 5
Number analyzed (Eyes) | 5
percentage change | -8.1 (14.6)

6. Secondary Outcome: Percentage Change in Retinal Thickness in the Study Eye at 12 Months Compared to Baseline
Description: Retinal thickness was assessed by spectral-domain optical coherence tomography (Cirrus HD-OCT; Carl Zeiss Meditec, Dublin, CA), a non-invasive imaging technique that uses long-wavelength light to capture micrometer-resolution cross-sectional images from biological tissue.
Time Frame: Baseline and 12 Months
Measure: Mean (Standard Deviation); unit: percentage change in retinal thickness
Units Other Than Participants: Eyes
Arm/Group | Minocycline
Number analyzed (Participants) | 3
Number analyzed (Eyes) | 3
percentage change in retinal thickness | -12.35 (1.21)

7. Secondary Outcome: Percentage Change in Retinal Thickness in the Study Eye at 18 Months Compared to Baseline
Description: as for outcome 6
Time Frame: Baseline and 18 Months
Measure: Mean (Standard Deviation); unit: percentage change in retinal thickness
Units Other Than Participants: Eyes
Arm/Group | Minocycline
Number analyzed (Participants) | 3
Number analyzed (Eyes) | 3
percentage change in retinal thickness | -20.09 (10.65)

8. Secondary Outcome: Percentage Change in Retinal Thickness in the Study Eye at 24 Months Compared to Baseline
Description: as for outcome 6
Time Frame: Baseline and 24 Months
Measure: Mean (Standard Deviation); unit: percentage change in retinal thickness
Units Other Than Participants: Eyes
Arm/Group | Minocycline
Number analyzed (Participants) | 3
Number analyzed (Eyes) | 3
percentage change in retinal thickness | -20.83 (4.62)

9. Secondary Outcome: Number of Study Eyes Demonstrating a Decrease in the Area of Late Leakage, as Measured by Fluorescein Angiography (FA), at 6 Months Compared to Baseline
Description: Fluorescein angiography (FA) images from both eyes in each participant were obtained via a standard digital imaging system (OIS, Sacramento, CA) at baseline and at Month 6, Month 12, Month 18, and Month 24. Three retinal specialists independently graded the area of late fluorescein leakage (at approximately 10 minutes)in each eye using a region-of-interest tool in an image analysis software package (NIH ImageJ, Bethesda, MD).
  The participant's eye that met the study eye eligibility criteria was selected as the study eye. For cases in which both eyes met the study eye eligibility criteria, the study eye was selected according to the "choice of study eye in cases of bilateral disease" selection criteria outlined in the eligibility criteria. The eye not chosen as the study eye is referred to as the "fellow eye."
Time Frame: 6 Months
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Minocycline
Number analyzed (Participants) | 5
Number analyzed (Eyes) | 5
Eyes | 5

10. Secondary Outcome: Number of Study Eyes Demonstrating a Decrease in the Area of Late Leakage, as Measured by Fluorescein Angiography (FA), at 12 Months Compared to Baseline
Description: as for outcome 9
Time Frame: 12 Months
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Minocycline
Number analyzed (Participants) | 3
Number analyzed (Eyes) | 3
Eyes | 3

11. Primary Outcome: Number of Study Eyes Demonstrating an Increase or Decrease in Best-corrected Visual Acuity (BCVA) of 15 or More Early Treatment Diabetic Retinopathy Study (ETDRS) Letters at 6 Months Compared to Baseline
Description: as for outcome 1
Time Frame: 6 months
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Minocycline
Number analyzed (Participants) | 5
Number analyzed (Eyes) | 5
Eyes | 1

12. Secondary Outcome: Number of Study Eyes Demonstrating a Decrease in the Area of Late Leakage, as Measured by Fluorescein Angiography (FA), at 18 Months Compared to Baseline
Description: as for outcome 9
Time Frame: 18 Months
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Minocycline
Number analyzed (Participants) | 3
Number analyzed (Eyes) | 3
Eyes | 3

13. Secondary Outcome: Number of Study Eyes Demonstrating a Decrease in the Area of Late Leakage, as Measured by Fluorescein Angiography (FA), at 24 Months Compared to Baseline
Description: as for outcome 9
Time Frame: 24 Months
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Minocycline
Number analyzed (Participants) | 3
Number analyzed (Eyes) | 3
Eyes | 3

14. Secondary Outcome: Number of Fellow Eyes Demonstrating a Decrease in the Area of Late Leakage, as Measured by Fluorescein Angiography (FA), at 6 Months Compared to Baseline
Description: as for outcome 9
Time Frame: 6 Months
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Minocycline
Number analyzed (Participants) | 5
Number analyzed (Eyes) | 5
Eyes | 4

15. Secondary Outcome: Number of Fellow Eyes Demonstrating a Decrease in the Area of Late Leakage, as Measured by Fluorescein Angiography (FA), at 12 Months Compared to Baseline
Description: as for outcome 9
Time Frame: 12 Months
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Minocycline
Number analyzed (Participants) | 3
Number analyzed (Eyes) | 3
Eyes | 1

16. Secondary Outcome: Number of Fellow Eyes Demonstrating a Decrease in the Area of Late Leakage, as Measured by Fluorescein Angiography (FA), at 18 Months Compared to Baseline
Description: as for outcome 9
Time Frame: 18 Months
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Minocycline
Number analyzed (Participants) | 3
Number analyzed (Eyes) | 3
Eyes | 2

17. Secondary Outcome: Number of Fellow Eyes Demonstrating a Decrease in the Area of Late Leakage, as Measured by Fluorescein Angiography (FA), at 24 Months Compared to Baseline
Description: as for outcome 9
Time Frame: 24 Months
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Minocycline
Number analyzed (Participants) | 3
Number analyzed (Eyes) | 3
Eyes | 1

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | Minocycline
Serious Adverse Events (participants affected / at risk) | 1/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Minocycline (N=6)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Minocycline (N=6)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Blepharitis (Eye disorders) | 1 (1)
Blood albumin decreased (Investigations) | 1 (1)
Blood glucose increased (Investigations) | 2 (2)
Blood magnesium decreased (Investigations) | 1 (1)
Blood thyroid stimulating hormone abnormal (Investigations) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (5)
Dizziness (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1)
Glycosylated haemoglobin increased (Investigations) | 1 (1)
Haemoglobin decreased (Investigations) | 2 (2)
Headache (Nervous system disorders) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Viral infection (Infections and infestations) | 1 (1)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1 (2)
White blood cell count increased (Investigations) | 1 (1)
Meibomianitis (Eye disorders) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1)
Tinea pedis (Infections and infestations) | 1 (1)
Blood pressure increased (Investigations) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (2)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No